CLINICAL TRIAL: NCT06065072
Title: Comparative Study of the Tomey OA-2000, Tomey CASIA2, and the LenStar LS900
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tomey Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Tomey OA-2000-001
Record Dates: First submitted 2023-09-12; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Cataract; Aphakic Eye; Pseudophakia
MeSH Terms: conditions — Cataract; Aphakia; Pseudophakia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Normal
  Interventions: Device: Optical measurement
- Cataract
  Interventions: Device: Optical measurement
- Special eye
  Interventions: Device: Optical measurement

INTERVENTIONS:
Device: Optical measurement — Optical measurements by optical biometers and an OCT

SUMMARY:
This is a prospective comparative study that will be conducted at one clinical site in the United States, in which subjects who sign an informed consent form and fulfil all inclusion and exclusion criteria, will have OCT scans obtained using the test and the predicate devices.

There will be two main types of analyses performed as part of this study, including 1) a precision analysis, and 2) an agreement analysis.

The precision analyses will be conducted utilizing all complete complements of acceptable scans from the test devices and predicate device for each of the 3 configurations. A complete complement of acceptable scans can be defined as subjects having 3 acceptable replicate scans on each of the 3 devices, at each of the 3 configurations. This is also synonymous with 3 scans for each of the 3 configurations on all 3 devices. If subjects have more than 3 acceptable scans per configuration on a device, only the first 3 will be considered for analyses.

The agreement analysis will be conducted utilizing the first set of acceptable scans from each instrument for all overlapping measurement types (for all measurement types two or more of the devices have in common) related to performance endpoints.

ELIGIBILITY:
Inclusion Criteria - Normal Cohort:

1. Male or female subjects 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study.

Inclusion Criteria - Cataract Cohort:

1. Male or female subjects 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study;
4. Subjects diagnosed with cataract classified per the LOCS III scale.

Inclusion Criteria - Special Eyes Cohort (eyes without a natural lens or eyes containing artificial materials):

1. Male or female subjects 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study;
4. Subjects diagnosed with one or both eyes having aphakia, pseudophakia or silicone oil.

Exclusion Criteria - Normal Cohort:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects who did not take off their contact lenses earlier than 15 minutes prior to the study;
3. Subjects with any current ocular pathology, as determined by self-report and confirmed by the investigator assessment and/or confirmed by the investigator assessment at the study visit;
4. Subjects that present with an active ocular infection in either eye;
5. Subjects who have a history of ocular surgery, including laser therapy/surgery;
6. Subjects with a condition or in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Exclusion Criteria - Cataract Cohort:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects who did not take off their contact lenses earlier than 15 minutes prior to the study;
3. Subjects with corneal or conjunctival abnormalities that may affect adequate assessment of the anterior chamber in either eye;
4. Subjects that present with an active ocular infection in either eye;
5. Subjects who have a history of ocular surgery, including laser therapy/surgery;
6. Subjects with a condition or in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Exclusion Criteria - Special Eyes Cohort (eyes without a natural lens or eyes containing artificial materials):

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects who did not take off their contact lenses earlier than 15 minutes prior to the study;
3. Subjects with corneal or conjunctival abnormalities that may affect adequate assessment of the anterior chamber in either eye;
4. Subjects that present with an active ocular infection in either eye;
5. Subjects with a condition or in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
6. Subjects with evidence of silicone oil emulsification;
7. Subjects with silicone oil in the anterior chamber;
8. Subjects with adherence of oil droplets to an intraocular lens.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal subjects (22 years of age or older) Cataract subjects (22 years of age or older), Special eyes subjects (22 years of age or older)
Sampling Method: Non-Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Agreement between the test devices and predicate device | Through study completion, approximately 4 months
  Agreement between each of the test devices and the predicate device will be evaluated by the mean difference and SD, the 95% limits of agreement (LOA), the Bland-Altman plots, and Deming regression for each subject population.
Precision of the test devices | Through study completion, approximately 4 months
  A crossed two-way random-effects analysis of variance (ANOVA) model will be used to estimate the repeatability and reproducibility limits of each scan parameter by subject population and study device (test and predicate device). This ANOVA model will include the configuration, subject, and interaction between configuration and subject as the factors. Repeatability and reproducibility standard deviations, as well as the corresponding coefficient of variations (CVs), will be calculated using this ANOVA model.
Safety of the test devices | Through study completion, approximately 4 months
  Adverse events reported will be listed by subject.

CONTACTS AND LOCATIONS:
Overall Officials: Ioanis Panagiotopoulos, Dr., Principal Investigator — NorthEast Eye Research Associates
Locations (1):
- NorthEast Eye Research Associates, Woburn, Massachusetts, United States